CLINICAL TRIAL: NCT02115334
Title: Development and Effectiveness of Home-based Programs for Preschool Children With Developmental Delay:a Randomized Controlled Trial.
Brief Title: Development and Effectiveness of Home-based Programs for Preschool Children With Developmental Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100-0996A3
Record Dates: First submitted 2013-09-27; First posted 2014-04-16 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2011-06

CONDITIONS: Developmental Delay
Keywords: Developmental delay; Early Intervention; Home programs; Preschool activities
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- professional-based group (Experimental): professional therapists delivering the PHPA
  Interventions: Behavioral: professional therapists delivering the PHPA
- parents-based group (Experimental): parents executing the PHPA
  Interventions: Behavioral: parents executing the PHPA
- control group (Active Comparator): health education only
  Interventions: Behavioral: health education

INTERVENTIONS:
Behavioral: professional therapists delivering the PHPA — PHPA are delivered by professional therapists, which including gross motor, fine motor, cognition verbal, social interactions, activity of daily living(ADL).
  Other Names: PHPA(delivered by professional therapists)
  Arms: professional-based group
Behavioral: parents executing the PHPA — PHPA are executed by parents, which including gross motor, fine motor, cognition verbal, social interactions, ADL.
  Other Names: PHPA (executed by parents)
  Arms: parents-based group
Behavioral: health education — health education of the children with DD.
  Arms: control group

SUMMARY:
Early intervention refers to the provision of early detection, early diagnosis, and early intervention for infants and young children with special needs. The implementation of home programs is very important for children with developmental delay (DD). Therefore, the purposes of this study are to: (1) design the preschool home program activities(PHPA), (2) investigate the immediate efficacy of PHPA for children with DD, (3) investigate the long-term efficacy of PHPA for children with DD.The second year is to investigate the immediate efficacy of PHPA for children with DD.

DETAILED DESCRIPTION:
A total of 36 children with DD, aged 2-6 years, were randomly assigned to the professional-based group (professional therapists delivering the PHPA, total n=13), parents-based group (parents executing the PHPA, n=12) and control group (health education only, n=11). Outcome measures included clinical assessments and subjective questionnaires. The clinical assessments were Comprehensive Developmental Inventory for Infants and Toddlers (CDIIT). The subjective questionnaires were Chinese Child Developmental Inventory (CCDI), Assessment of preschool children's participation (APCP), TN0-AZL Preschool quality of life (TAPQOL) and parent stress index (PSI). Tests were administrated before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 6-years-old children
* clinical diagnosis of DD and other related disorders

Exclusion Criteria:

* unstable physiological conditions
* progression or regression symptoms

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in clinical assessment after 8 weeks intervention of PHPA at 6 months | baseline, 8 weeks, 3 months, 6 months
  The clinical assessments were Comprehensive Developmental Inventory for Infants and Toddlers (CDIIT).

SECONDARY OUTCOMES:
change from baseline in Chinese Child Developmental Inventory (CCDI) after 8 weeks intervention of PHPA at 6 months | baseline, 8 weeks, 3 months, 6 months
  Measurement of CCDI.
change from baseline in Assessment of preschool children's participation(APCP) after 8 weeks intervention of PHPA at 6 months | baseline, 8 weeks, 3 months, 6 months
  Measurement of APCP.
change from baseline in TN0-AZL Preschool quality of life (TAPQOL) after 8 weeks intervention of PHPA at 6 months | baseline, 8 weeks, 3 months, 6 months
  Measurement of TAPQOL.
change from baseline in parent stress index (PSI) after 8 weeks intervention of PHPA at 6 months | baseline, 8 weeks, 3 months, 6 months
  Measurement of PSI.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD,PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taoyuan, Taiwan